CLINICAL TRIAL: NCT00925717
Title: of PATient Education Related to CV Risk factOrs in Type 2 Diabetes Mellitus(Patrol).
Acronym: DART
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Hyunah Caroline, Choi / CV TA Physician, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CKR-DUM-2009/1
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Low Density Lipoprotein Cholesterol Goal Achievement
Keywords: ADA recommendation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 2500 patients: Who have records of clinic visit with endocrine internal medicines of nationwide secondary/tertiary hospitals within the last six months.

SUMMARY:
An observational, non-interventional, multi-centre study to provide further information on the utility of test for a predictive marker by investigating the current prevalence of high sensitivity CRP (hs-CRP) testing and characteristics of each CVD risk group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who was diagnosed as diabetes
* Subjects who was diagnosed as dyslipidaemia or takes lipid lowering medication
* Clinic visit in the past 6 months more than once

Exclusion Criteria:

* Subjects who are unwilling or unable to provide their examination and lab result of medical chart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Who have records of clinic visit with endocrine internal medicines of nationwide secondary/tertiary hospitals within the last six months.
Sampling Method: Non-Probability Sample
Enrollment: 4045 (Actual)
Dates: Start 2009-05; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Investigate LDL-C goal achievement rate according to ADA recommendation | Within the last 6 months from the date of data entry.

SECONDARY OUTCOMES:
Investigate reduction of 10-year risk for CHD by using UKPDS risk engine | Within the last 6 months from the date of data entry.

CONTACTS AND LOCATIONS:
Overall Officials: MoonGyu Lee, Ph.D., Study Director — Samsung Medical Center
Locations (22):
- South Korea (22):
  - Research Site, Cheonan-si, Chungchungnam-do
  - Research Site, Chuncheon, Gangwon-do
  - Research Site, Gangneung, Gangwon-do
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Ansan-si, Gyeonggi-do
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Uijeongbu-si, Gyeonggi-do
  - Research Site, Gwangju-si, Jeollanam-do
  - Research Site, Suncheon, Jeollanam-do
  - Research Site, Jeonju, Jeonllabuk-do
  - Research Site, Busan
  - Research Site, Cheonju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Kwangju-si
  - Research Site, Seoul